# Reducing Disparities in Access to Kidney Transplantation: the RaDIANT Regional Study

NCT02389387

Date: 11/19/2020

### Emory University Verbal Consent to be a Research Subject / HIPAA Authorization

**<u>Title</u>**: Evaluation of RaDIANT Regional Study

Principal Investigator: Rachel Patzer, PhD, MPH

**Sponsor:** National Institutes of Health

#### Introduction

We are conducting a study to evaluate interventions that were conducted in dialysis facilities. It is entirely your choice whether or not to participate. If you decide to take part, you can change your mind later on and leave the research study. The decision to join or not join the research study will not cause you to lose any medical benefits. If you decide not to take part in this study, your doctor will continue to treat you.

#### What is the purpose of this study?

The purpose of this study is to evaluate the interventions conducted in your dialysis facility. You will be asked to complete a survey to help us understand your experience with these interventions.

We would like to know if you would be interested in completing a brief phone survey. This survey will take a maximum of 15 minutes to complete. Your answers will be shared with Emory researchers, but we will not record your name when recording your answers. The survey will ask you about your experience with different educational materials, including a patient video.

#### **Risks and Benefits**

As a participant in this study, the only risk to you is to your privacy. To protect your privacy, we will follow federal and state privacy laws, including the Health Insurance Portability and Accountability Act (or, HIPAA) and will not record your name.

This study may not benefit you directly, but we hope this research will help us plan ways to help other patients in the future have better health care.

#### Compensation

You will receive a \$10 gift card to thank you for your participation and time. There are no costs to you associated with the study.

#### **Protection of Private Information**

Your privacy is very important to us. Your health information that identifies you is your "protected health information" (PHI). To protect your PHI, we will follow federal and state privacy laws, including the Health Insurance Portability and Accountability Act (HIPAA).

Whenever possible, a study number, rather than your name, will be used on study records. Your name and other identifying information will not appear when we present or publish the study results.

The following persons or groups may use your PHI for this study: The Principal Investigator and the research staff

Page 1 of 3 IRB Form 07202015 Version Date: 01/07/2016

### Emory University IRB IRB use only

Document Approved On: «ApproveDate»

Version Date: 01/07/2016

- National Institutes of Health, Network 6, and people or companies they use to carry out the study
- Emory offices who are part of the Human Research Participant Protection Program, and those who are involved in research-related administration and billing
- Any government agencies who regulate the research including the Office for Human Research Protections (OHRP)
- Any other parties that apply including possible future researchers who want to contact subjects for studies

We will disclose your PHI when required to do so by law in addition to subpoenas or court orders.

You may revoke your authorization at any time by calling or writing the Principal Investigator:



If identifiers (like your name, address, and telephone number) are removed from your PHI, then the remaining information will not be subject to the Privacy Rules. This means that the information may be used or shared with other people or organizations, and/or for other purposes.

If we share your PHI with other groups who do not have to follow the Privacy Rule, then they could use or share your PHI to others without your authorization. Your authorization will not expire because your PHI will need to be kept indefinitely for research purposes. Let me know if you have questions about this

#### **Contact Information**

If you have questions about this study, your part in it, your rights as a research participant, or if you have questions, concerns or complaints about the research you may contact the following:

| Rachel Patzer, PhD, Principal Inves | igator, at |
|-------------------------------------|------------|
| Emory Institutional Review Board: | |

IRB00079596 IRB Approved 11/19/2020 Study No.: «ID»

## Emory University IRB IRB use only

Document Approved On: «ApproveDate»

Version Date: 01/07/2016

| Consen | ĺ |
|--------|---|
|--------|---|

| Do you have any questions about any | thing I just s | aid? Were there any | parts that seemed ur | nclear? |
|---|---|---|---|---|
| Do you agree to take part in the study | <b>/</b> ? | | | |
| Participant agrees to participate: | Yes | No | | |
| If Yes: | | | | |
| Name of Participant | | | _ | |
| Signature of Person Conducting Informed Consent Discussion | | | Date | Time |
| Name of Person Conducting Informed | d Consent Dis | scussion | _ | |